CLINICAL TRIAL: NCT05754008
Title: A Randomized Trial of Care Navigator to Support Younger Latinx Adults Newly Diagnosed With Type 2 Diabetes (AURORA)
Brief Title: Care Navigator Support for Younger Latinx Adults With Type 2 Diabetes
Acronym: AURORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1833646
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Care Navigator, Latinx
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study team will conduct a patient-level randomized, parallel-group pragmatic trial of usual care vs. the AURORA care strategy among Latinx members (ages 18-44), recently diagnosed with T2D with a diagnosis HbA1c ≥8% (n=102/study arm). Outcomes assessed at 6 months post-enrollment will include HbA1c changes, medication initiation and adherence, and changes in patient-reported measures (e.g., self-efficacy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AURORA Care Strategy (Experimental): Participants will receive the AURORA Care Strategy in addition to their usual diabetes care.
  Interventions: Behavioral: AURORA Care Strategy
- Usual Care (No Intervention): No intervention will be employed. This arm will continue to receive their usual diabetes care.

INTERVENTIONS:
Behavioral: AURORA Care Strategy — Participants will be invited to partake in three telemedicine visits with the care navigator during the months following diagnosis. The visits center around proactive and tailored T2D self-management support.
  Arms: AURORA Care Strategy

SUMMARY:
The study proposes to rigorously evaluate a proactive, culturally responsive care navigator intervention targeting younger-onset Latinx individuals with a new T2D diagnosis (AURORA [Active Outreach to Younger Latinx]) within Kaiser Permanente Northern California (KPNC).

DETAILED DESCRIPTION:
The study has three primary objectives: 1) learn what is required to create and sustain a care navigator workforce and document our experience hiring a care navigator for the study, 2) implement and evaluate the AURORA strategy within KPNC, and 3) refine and adapt the AURORA strategy for future Kaiser Permanente (KP) wide dissemination. The AURORA strategy centers on a care navigator who will proactively conduct three telemedicine visits tailored to Latinx adults with early onset type 2 diabetes (T2D, defined as age <45 years). The AURORA strategy will conducted with the following five goals: 1) assessment of familiarity and use of T2D care within KP, 2) assessment of individual's self-management support needs, 3) motivational interviewing to support behavior change, 4) pragmatic skills training, including use of crucial technologies to support self-management, and 5) matching member's needs with existing KPNC T2D resources.

ELIGIBILITY:
Inclusion Criteria:

* KPNC member, age >20 and age <45 with
* New clinical diagnosis of T2D within the prior 1-8 months
* HbA1c≥8%. If the study team are having trouble recruiting an adequate sample, the study team may lower the HbA1c threshold to ≥7.5%
* Proficient (written and spoken) in English or Spanish

Exclusion Criteria:

* Pregnant women
* Type 1 Diabetes

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differences between study arms in HbA1c change 6-months following enrollment | 6-months following enrollment
  Change in HbA1c will be assessed using HbA1c values obtained through routine care, with the most recent HbA1c preceding study enrollment and the HbA1c value closest to 6-months following enrollment used to assess HbA1c change.

SECONDARY OUTCOMES:
Healthcare contact | 6-months following enrollment
  Differences in healthcare contact with members of the T2D diabetes care team, including care manager, PCPs, educators.
Completion of recommended HbA1c monitoring | 6-months following enrollment
  Completing HbA1c labs
T2D-related medication initiation | 6-months following enrollment
  Initiation of T2D-related medication
T2D-related medication adherence | 6-months following enrollment
  Adherence to T2D-related medication
Use of remote glucose monitoring to measure glucose levels | 6-months following enrollment
  Use of a remote glucose monitoring to measure glucose levels
Participant-reported measures: Confidence in Accessing Care | 3-months following enrollment
  Assessed at 3-month survey
Participant-reported measures: Diet and Exercise | 3-months following enrollment
  Assessed at 3-month survey
Participant-reported measures: Self-efficacy for diabetes | 3-months following enrollment
  Assessed at 3-month survey
Participant-reported measures: Motivation and locus of control | 3-months following enrollment
  Assessed at 3-month survey
Participant-reported measures: Diabetes distress | 3-months following enrollment
  Assessed at 3-month survey
Participant-reported measures: Diabetes stigma | 3-months following enrollment
  Assessed at 3-month survey

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Gopalan, MD, MS, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilmot E, Idris I. Early onset type 2 diabetes: risk factors, clinical impact and management. Ther Adv Chronic Dis. 2014 Nov;5(6):234-44. doi: 10.1177/2040622314548679. PMID 25364491
- [Background] Gopalan A, Mishra P, Alexeeff SE, Blatchins MA, Kim E, Man A, Karter AJ, Grant RW. Initial Glycemic Control and Care Among Younger Adults Diagnosed With Type 2 Diabetes. Diabetes Care. 2020 May;43(5):975-981. doi: 10.2337/dc19-1380. Epub 2020 Mar 4. PMID 32132007
- [Background] Laiteerapong N, Ham SA, Gao Y, Moffet HH, Liu JY, Huang ES, Karter AJ. The Legacy Effect in Type 2 Diabetes: Impact of Early Glycemic Control on Future Complications (The Diabetes & Aging Study). Diabetes Care. 2019 Mar;42(3):416-426. doi: 10.2337/dc17-1144. Epub 2018 Aug 13. PMID 30104301
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] American Diabetes Association. 1. Improving Care and Promoting Health in Populations: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S7-S14. doi: 10.2337/dc21-S001. PMID 33298412
- [Background] Hildebrand JA, Billimek J, Lee JA, Sorkin DH, Olshansky EF, Clancy SL, Evangelista LS. Effect of diabetes self-management education on glycemic control in Latino adults with type 2 diabetes: A systematic review and meta-analysis. Patient Educ Couns. 2020 Feb;103(2):266-275. doi: 10.1016/j.pec.2019.09.009. Epub 2019 Sep 9. PMID 31542186
- [Background] Flores-Luevano S, Pacheco M, Shokar GS, Dwivedi AK, Shokar NK. Impact of a Culturally Tailored Diabetes Education and Empowerment Program in a Mexican American Population Along the US/Mexico Border: A Pragmatic Study. J Clin Med Res. 2020 Aug;12(8):517-529. doi: 10.14740/jocmr4273. Epub 2020 Jul 22. PMID 32849940
- [Background] Rosal MC, Ockene IS, Restrepo A, White MJ, Borg A, Olendzki B, Scavron J, Candib L, Welch G, Reed G. Randomized trial of a literacy-sensitive, culturally tailored diabetes self-management intervention for low-income latinos: latinos en control. Diabetes Care. 2011 Apr;34(4):838-44. doi: 10.2337/dc10-1981. Epub 2011 Mar 4. PMID 21378213
- [Background] Islam NS, Wyatt LC, Taher MD, Riley L, Tandon SD, Tanner M, Mukherji BR, Trinh-Shevrin C. A Culturally Tailored Community Health Worker Intervention Leads to Improvement in Patient-Centered Outcomes for Immigrant Patients With Type 2 Diabetes. Clin Diabetes. 2018 Apr;36(2):100-111. doi: 10.2337/cd17-0068. PMID 29686448
- [Background] Spencer MS, Gunter KE, Palmisano G. Community health workers and their value to social work. Soc Work. 2010 Apr;55(2):169-80. doi: 10.1093/sw/55.2.169. PMID 20408358
- [Background] Hartzler AL, Tuzzio L, Hsu C, Wagner EH. Roles and Functions of Community Health Workers in Primary Care. Ann Fam Med. 2018 May;16(3):240-245. doi: 10.1370/afm.2208. PMID 29760028
- [Background] Adair R, Wholey DR, Christianson J, White KM, Britt H, Lee S. Improving chronic disease care by adding laypersons to the primary care team: a parallel randomized trial. Ann Intern Med. 2013 Aug 6;159(3):176-84. doi: 10.7326/0003-4819-159-3-201308060-00007. PMID 23922063
- [Background] Palmas W, March D, Darakjy S, Findley SE, Teresi J, Carrasquillo O, Luchsinger JA. Community Health Worker Interventions to Improve Glycemic Control in People with Diabetes: A Systematic Review and Meta-Analysis. J Gen Intern Med. 2015 Jul;30(7):1004-12. doi: 10.1007/s11606-015-3247-0. Epub 2015 Mar 4. PMID 25735938
- [Background] Kvedar J, Coye MJ, Everett W. Connected health: a review of technologies and strategies to improve patient care with telemedicine and telehealth. Health Aff (Millwood). 2014 Feb;33(2):194-9. doi: 10.1377/hlthaff.2013.0992. PMID 24493760
- [Background] Ray KN, Chari AV, Engberg J, Bertolet M, Mehrotra A. Disparities in Time Spent Seeking Medical Care in the United States. JAMA Intern Med. 2015 Dec;175(12):1983-6. doi: 10.1001/jamainternmed.2015.4468. No abstract available. PMID 26437386
- [Background] Reed ME, Huang J, Parikh R, Millman A, Ballard DW, Barr I, Wargon C. Patient-Provider Video Telemedicine Integrated With Clinical Care: Patient Experiences. Ann Intern Med. 2019 Aug 6;171(3):222-224. doi: 10.7326/M18-3081. Epub 2019 Apr 30. No abstract available. PMID 31035294
- [Background] Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998 Aug-Sep;1(1):2-4. No abstract available. PMID 10345255
- [Background] Wan EYF, Fung CSC, Jiao FF, Yu EYT, Chin WY, Fong DYT, Wong CKH, Chan AKC, Chan KHY, Kwok RLP, Lam CLK. Five-Year Effectiveness of the Multidisciplinary Risk Assessment and Management Programme-Diabetes Mellitus (RAMP-DM) on Diabetes-Related Complications and Health Service Uses-A Population-Based and Propensity-Matched Cohort Study. Diabetes Care. 2018 Jan;41(1):49-59. doi: 10.2337/dc17-0426. Epub 2017 Nov 14. PMID 29138274
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Background] Gopalan A, Blatchins MA, Altschuler A, Mishra P, Fakhouri I, Grant RW. Disclosure of New Type 2 Diabetes Diagnoses to Younger Adults: a Qualitative Study. J Gen Intern Med. 2021 Jun;36(6):1622-1628. doi: 10.1007/s11606-020-06481-y. Epub 2021 Jan 26. PMID 33501523
- [Background] Klompas M, Eggleston E, McVetta J, Lazarus R, Li L, Platt R. Automated detection and classification of type 1 versus type 2 diabetes using electronic health record data. Diabetes Care. 2013 Apr;36(4):914-21. doi: 10.2337/dc12-0964. Epub 2012 Nov 27. PMID 23193215
- [Background] Makam AN, Nguyen OK, Moore B, Ma Y, Amarasingham R. Identifying patients with diabetes and the earliest date of diagnosis in real time: an electronic health record case-finding algorithm. BMC Med Inform Decis Mak. 2013 Aug 1;13:81. doi: 10.1186/1472-6947-13-81. PMID 23915139
- [Background] Pandit AU, Bailey SC, Curtis LM, Seligman HK, Davis TC, Parker RM, Schillinger D, DeWalt D, Fleming D, Mohr DC, Wolf MS. Disease-related distress, self-care and clinical outcomes among low-income patients with diabetes. J Epidemiol Community Health. 2014 Jun;68(6):557-64. doi: 10.1136/jech-2013-203063. Epub 2014 Jan 31. PMID 24489044
- [Background] Ratanawongsa N, Karter AJ, Parker MM, Lyles CR, Heisler M, Moffet HH, Adler N, Warton EM, Schillinger D. Communication and medication refill adherence: the Diabetes Study of Northern California. JAMA Intern Med. 2013 Feb 11;173(3):210-8. doi: 10.1001/jamainternmed.2013.1216. PMID 23277199
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Molyneaux LM, Constantino MI, McGill M, Zilkens R, Yue DK. Better glycaemic control and risk reduction of diabetic complications in Type 2 diabetes: comparison with the DCCT. Diabetes Res Clin Pract. 1998 Nov;42(2):77-83. doi: 10.1016/s0168-8227(98)00095-3. PMID 9886743
- [Background] The relationship of glycemic exposure (HbA1c) to the risk of development and progression of retinopathy in the diabetes control and complications trial. Diabetes. 1995 Aug;44(8):968-83. PMID 7622004
- [Background] White IR, Royston P, Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. Stat Med. 2011 Feb 20;30(4):377-99. doi: 10.1002/sim.4067. Epub 2010 Nov 30. PMID 21225900
- [Background] Rubin DB, Schenker N. Multiple imputation in health-care databases: an overview and some applications. Stat Med. 1991 Apr;10(4):585-98. doi: 10.1002/sim.4780100410. PMID 2057657
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Barbosa CE, Masho SW, Carlyle KE, Mosavel M. Factors Distinguishing Positive Deviance Among Low-Income African American Women: A Qualitative Study on Infant Feeding. J Hum Lact. 2017 May;33(2):368-378. doi: 10.1177/0890334416673048. Epub 2016 Nov 24. PMID 27881731
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol 2006;3(2):77-101. DOI: 10.1191/1478088706qp063oa.